CLINICAL TRIAL: NCT01003899
Title: A Phase II Trial of BIBW 2992 as a Third-line Treatment for Patients With Stage IIIB/IV Adenocarcinoma of the Lung Harbouring Wild-type EGFR
Brief Title: A Phase II Trial of Afatinib(BIBW 2992) in Third-line Treatment for Patients With Stage IIIB/IV Adenocarcinoma of the Lung Harbouring Wild-type Epidermal Growth Factor Receptor[EGFR]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.72
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Results first posted 2013-10-17 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- afatinib (BIBW 2992) (Experimental): patient to receive afatinib(BIBW 2992) po QD in an open-label manner
  Interventions: Drug: afatinib (BIBW 2992)

INTERVENTIONS:
Drug: afatinib (BIBW 2992) — afatinib (BIBW 2992) po QD

SUMMARY:
To explore the efficacy of BIBW 2992 defined by the objective response rate (Complete Response, Partial Response) as determined by Response Evaluation Criteria in Solid Tumours[RECIST] 1.1 in the patients with advanced (stage IIIB or IV) adenocarcinoma of the lung harbouring wild-type EGFR.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically confirmed stage IIIB/IV adenocarcinoma in non-small cell lung cancer[NSCLC]
2. Progressive disease following a second-line cytotoxic chemotherapy including at least one platinum-containing regimen
3. A known wild-type EGFR status
4. Patients 18 years of age or older

Exclusion criteria:

1. More than two prior cytotoxic chemotherapy treatment regimens for relapsed or metastatic disease
2. Prior treatment with EGFR targeting small molecules or antibodies
3. Radiotherapy or surgery within 4 weeks prior to study entry
4. Active brain metastasis
5. Known pre-existing interstitial lung disease
6. History or presence of clinically relevant cardiovascular abnormalities
7. Cardiac left ventricular function with resting ejection fraction of less than 50%
8. Absolute neutrophil count[ANC] < 1,500/mm3
9. Platelet count <100,000/mm3
10. Creatinine clearance<60ml/min or serum creatinine >1.5 times upper limit of normal
11. Women of childbearing potential, or men who are able to father a child, unwilling to use a medically acceptable method of contraception during the trial
12. Pregnancy or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- South Korea (3):
  - 1200.72.8201 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.72.8202 Boehringer Ingelheim Investigational Site, Seoul
  - 1200.72.8203 Boehringer Ingelheim Investigational Site, Seoul

REFERENCES:
- [Derived] Ahn MJ, Kim SW, Cho BC, Ahn JS, Lee DH, Sun JM, Massey D, Kim M, Shi Y, Park K. Phase II study of Afatinib as third-line treatment for patients in Korea with stage IIIB/IV non-small cell lung cancer harboring wild-type EGFR. Oncologist. 2014 Jul;19(7):702-3. doi: 10.1634/theoncologist.2013-0419. Epub 2014 May 27. PMID 24868099

RESULTS

PARTICIPANT FLOW:
Groups:
- Afatinib 40 mg: Afatinib 40 mg film coated tablets where administered on continuous daily dosing until progression, unacceptable adverse events or other reasons necessitating withdrawal
Period: Overall Study
Arm/Group | Afatinib 40 mg
Started | 47 (enrolled)
Completed | 0
Not Completed | 47
Not completed — Other Adverse Event | 8
Not completed — Not entered | 4
Not completed — Not treated | 1
Not completed — Progressive disease | 34

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) consists of all patients treated with at least one dose of study drug.
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Best Objective Response
Description: Percentage of participants with best objective response: confirmed complete response (CR) or confirmed partial response (PR) according to RECIST (version 1.1).
Time Frame: Baseline till progression or death
Population: FAS (Full Analysis Set). The FAS consisted of all treated patients, excluding any patients found not be EGFR mutation negative according to central laboratory testing.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 38
Percentage of participants | 0 [0 to 9]

2. Secondary Outcome: Percentage of Participants With Disease Control (DC)
Description: Percentage of participants with objective response or stable disease (SD) as determined by RECIST version 1.1.
Time Frame: Baseline till progression or death
Population: FAS - Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 38
Percentage of participants | 24 [11 to 40]

3. Secondary Outcome: Progression Free Survival (PFS) Time
Description: PFS time is defined as time from start of treatment to the earliest of progression (RECIST version 1.1), clinical progression (investigator), start of new anti-cancer treatment or death
Time Frame: Baseline till end of study or death
Population: FAS - Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 38
Weeks | 4.07 ((11, 40)) [3.86 to 8.00]

4. Secondary Outcome: Duration of Disease Control (DC)
Description: Duration of diesease control (DC) (objective response or stable disease (SD) as determined by RECIST version 1.1).
Time Frame: Baseline till progression or death
Population: FAS - Full Analysis Set
Measure: Median (Full Range); unit: weeks
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 9
weeks | 19.29 [11.6 to 43.1]

5. Secondary Outcome: Time to OR
Description: The time to objective response (OR) was the duration from the first treatment to the time when the measurement criteria for CR and/or PR were met according to RECIST 1.1 criteria.
Time Frame: Baseline till progression or death
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of OR
Description: Duration of OR was measured from the time the criteria for CR or PR (whichever was documented first) were first met until the first date that progressive disease or death was objectively documented.
Time Frame: Baseline till progression or death
Arm/Group | Afatinib 40 mg
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | Afatinib 40 mg
Serious Adverse Events (participants affected / at risk) | 17/42
Other Adverse Events (participants affected / at risk) | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=42)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 5
Blood creatinine increased (Investigations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg (N=42)
Abdominal pain (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 26
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 3
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 5
Fatigue (General disorders) | 4
Mucosal inflammation (General disorders) | 12
Pyrexia (General disorders) | 3
Paronychia (Infections and infestations) | 13
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 18
Back pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Acne (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 7
Nail disorder (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 32
Skin exfoliation (Skin and subcutaneous tissue disorders) | 6
Skin fissures (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.